CLINICAL TRIAL: NCT04822389
Title: Effect of the Physical Exercise Training Using Telerehabilitation Among Lymphoma Patients: A Pilot Study
Brief Title: Telerehabilitation and Lymphoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IPRHO-KOREHAB2021
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Lymphoma; Rehabilitation
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based telerehabilitation exercise (Experimental): Exercise training is conducted in the patient's home conditions using modern technology to transfer medical data remotely - the participants receive a heart rate monitor and sensor. To know what to do and how to exercise, the first (1-2) exercise training sessions will be controlled by the physiotherapist in a rehabilitation clinic in the hospital, who creates individual exercise training for each patient. The patient's training data will be downloaded and updated regularly via the internet platform and clinicians will evaluate these results and provide patients with telephone feedback.
  Interventions: Device: Telerehablitation using heart rate monitor

INTERVENTIONS:
Device: Telerehablitation using heart rate monitor — Eligible participants will undergo 12 weeks of physical exercise using a heart rate monitor and internet platform at home. The participants will regularly (minimum once per week) upload the exercise data from the heart rate monitor into the internet platform. An exercise telerehabilitation session consists of the warm-up phase, aerobic phase (30 - 50 minutes gradually increasing exercise duration; heart rate zone based on baseline cardiopulmonary exercise test) and cool-down phase. The exercise training period is set to 3 times a week for 12 weeks. Study participants will receive user guides developed by research team with detailed instructions regarding equipment set-up, training protocol, and contact information. Also, participants will receive weekly phone calls from week 0 to week 12 to monitor adverse events, encourage compliance and adherence to the study protocol, address any subject questions or concerns, and collect information regarding participants' current symptomatology.

SUMMARY:
This study aims to examine the feasibility and effect of a home-based short-term telerehabilitation exercise intervention using heart rate monitor and internet platform in patients with lymphoma.

DETAILED DESCRIPTION:
Fifteen lymphoma cancer patients post-treatment (except adjuvant treatment) will be enrolled in the study. Cardiorespiratory fitness (peak oxygen consumption), adverse events, body composition and adherence to exercise prescription will be evaluated at baseline, 12-week, and year after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Lymphoma patients post-treatment (except ongoing adjuvant treatment)
* Post-treatment period not exceeding 3 months
* Internet connection at home
* Literacy with information and communication technology
* Patients who agreed with informed consent

Exclusion Criteria:

* Inability to perform a cardiopulmonary exercise test
* Psychological severe or cognitive disorders
* Contraindications for cardiopulmonary exercise testing
* Other exercise limitations (musculoskeletal disorders)
* Planned intervention or operation
* Participants who are enrolled in or participate in other rehabilitation program
* Participants who plan to be or are included in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (CRF) | Change from baseline to 12 weeks and 1-year
  Peak oxygen uptake (VO2peak) during the cardiopulmonary exercise test

SECONDARY OUTCOMES:
Body composition (Total muscle mass in kilograms) | Change from baseline to 12 weeks and 1-year
  Total muscle mass is the amount of muscle in body, including skeletal muscles, smooth muscles, and cardiac muscles. Total muscle mass will be measured by bioelectrical impedance analysis.
Body composition (Body fat mass in kilograms) | Change from baseline to 12 weeks and 1-year
  Body fat mass is the actual weight of fat in body. Body fat mass will be measured by bioelectrical impedance analysis.
Body composition (Body weight in kilograms) | Change from baseline to 12 weeks and 1-year
  Body weight is the measurement of weight without items located on the person. Body weight will be measured by bioelectrical impedance analysis.
Incidence of treatment-emergent adverse events assessed by 5 grade scale | Data will be recorded continuously from the baseline to 12 weeks
  Participants will be encouraged to use the contact details for reporting the incidence of treatment-emergent adverse events at any time throughout the study period. The type, incidence, and severity of adverse events by scale (Grade 1: Mild, asymptomatic or mild symptoms; Grade 2: Moderate, minimal; Grade 3: Severe or medically significant; Grade 4: Life-threatening consequences; and Grade 5: Death) will be noted
Exercise adherence | 12 weeks
  Exercise adherence is defined as number of exercise sessions attended of a possible 36 offered by the exercise intervention program. Exercise adherence will be determined by participant exercise web datasheet review at 12 weeks.
Exercise compliance | 12 weeks
  Number of participants who attend atleast 70% of prescribed exercise sessions measured by exercise datasheet at 12 weeks. (70% of prescribed exercise sessions = 25 exercise sessions in 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ladislav Batalik, Principal Investigator — Department of Rehabilitation, University Hospital Brno, Czech Republic
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Filakova K, Janikova A, Felsoci M, Dosbaba F, Su JJ, Pepera G, Batalik L. Home-based cardio-oncology rehabilitation using a telerehabilitation platform in hematological cancer survivors: a feasibility study. BMC Sports Sci Med Rehabil. 2023 Mar 23;15(1):38. doi: 10.1186/s13102-023-00650-2. PMID 36959613